CLINICAL TRIAL: NCT02271815
Title: A Clinical and Imaging Study to Evaluate a Novel Dentifrice
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Livionex Inc. (Industry)
Responsible Party: Principal Investigator, Petra E. Wilder-Smith, Professor, Director of Dentistry, University of California, Irvine
Other Study IDs: 20139778; Livionex, Inc. (Other: Livionex, Inc.)
Record Dates: First submitted 2014-10-09; First posted 2014-10-22 (Estimated); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Gingivitis; Periodontitis; Dental Plaque
Keywords: toothpaste; dental gel; dentifrice; plaque removal; oral biofilm; plaque accumulation
MeSH Terms: conditions — Gingivitis; Periodontitis; Dental Plaque | interventions — Oral Hygiene

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral Hygiene: Oral Hygiene
  Interventions: Other: Oral Hygiene

INTERVENTIONS:
Other: Oral Hygiene — Oral Hygiene

SUMMARY:
There is a need for toothpastes that more effectively remove oral biofilm, inhibit biofilm re-formation and support periodontal health. This is particularly important for patients with long-term orthodontic fixtures or prosthodontic appliances, and also for debilitated, diabetic and immunocompromised patients. The objective of this study is to evaluate the effects of toothpastes on plaque presence and removal, gingival and periodontal health, dental hard tissue mineralization, erosion, abrasion, and microstructure as well as dry/sore mouth. In addition to clinical scoring and photographs, tooth and gum sensitivity, saliva volume, pH and buffering and enamel health may be evaluated using tooth samples worn on removable dental retainers. These samples will be examined outside of the mouth using advanced optical techniques such as Optical Coherence Tomography (OCT), Fluorescence, various forms of microscopy and spectroscopy.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the in vivo effects of toothpastes and dental gels on gingival and periodontal health, enamel demineralization, remineralization and microstructure . The purpose of this study is to evaluate the effects of over-the-counter toothpastes and dental gels including Colgate Total, Crest Cavity Protection, Zendium Classic toothpaste, and Livionex LivFree and LivFresh using established clinical evaluation parameters as well as innovative imaging approaches (Optical Coherence Tomography and Multiphoton Microscopy) to measure the status of the oral tissues

Imaging devices:

* Optical Coherence Tomography can be used to identify and measure inflammation of the gums and gum pockets.The results can be used to evaluate the health of the gums, and changes caused by using specific toothpastes
* Multiphoton Microscopy can be used to identify and measure bacterial plaque or biofilm in the mouth. The results can determine effects of specific toothpastes on the development and breakup of bacterial biofilm or plaque.

In the first part of this study, subjects with moderate gingival inflammation (Löe and Silness Gingival Index ≥2) and pocket depths <4 will be randomly assigned to brush twice daily for 21 days with the test or the control dental gel. On Days 0, 7, 14, and 21, plaque levels (Quigley-Hein, Turesky Modification Plaque Index), gingival inflammation (Löe and Silness Gingival Index), and gingival bleeding (modified Sulcus Bleeding Index) will be determined by one blinded, investigator (Dr. Wilder-Smith) using standard probing techniques. In vivo Optical Coherence Tomography (OCT) and Multiphoton Microscopy (MPM) will be used for in situ imaging. The results from this study will help evaluate the effects of the test dentifrice formulation on plaque removal and maintaining gingival health.

In the second part of this study, plaque formation and removal will be quantified in subjects using ex vivo Optical Coherence Tomography (OCT) and Multiphoton Microscopy (MPM) imaging of small enamel chips mounted on a simple intra-oral retainer. In this cross-over design study, the subjects will attend the test site on 11 occasions over an 11-week period. Subjects will have an intra-oral retainer manufactured, which will be worn for a minimum of 22 hours per day and will have up to 8 sterile human enamel inserts fitted.This study will be conducted in three arms with a maximum of 44h of retainer wear during each arm, and each study arm will follow the same procedure. 2 different over-the-counter toothpastes and a water control will be used for each arm of the study, respectively. There will be a minimum of two weeks between each study arm.

The third part of this study will involve subjects with no specific oral health issues. The protocol will involve subjects wearing simple retainers for 3 periods of 2 weeks each with 5 sterilized enamel chips attached in the palate area. The study will have 3 arms using a control and 2 active toothpastes. There will be washout of 1-2 weeks between each study arm. Samples will be analyzed outside of the mouth using OCT and MPM techniques, as well as micro computer tomography (microCT), Energy Dispersive Spectroscopy (EDS) and X-Ray Photoelectron Spectroscopy (XPS). (Section 3 has been completed as of July 11, 2016)

The fourth part of this study will involve subjects with xerostomia. Subjects will wear simple removable retainers for 2 periods of 1 week each, with 5 sterilized demineralized enamel chips attached in the palate area of the retainer. Fresh enamel chips will be used for each arm of the study. After study completion, chips will be used for Scanning Electron microscopy (SEM) and microhardness measurement. We will provide custom retainers made from impressions of each subject. Upon conclusion of the study, we will analyze the effects of each toothpaste on surface enamel using scanning electron microscopy (SEM) and microhardness as well as microCT, EDS and XPS data.

In the fifth part of this study, plaque formation and removal in subjects will be quantified using the standard clinical index for plaque levels (Quigley-Hein, Turesky Modification Plaque Index). This will be determined by one blinded investigator using a periodontal probe. In addition, ex vivo Optical Coherence Tomography (OCT) and Multiphoton Microscopy (MPM) imaging of biofilm samples will be performed on plaque specimens collected using standardized technique and a 2mm curette. In this 3-arm cross-over double-blinded study, the subjects will attend the test site for up to 7 occasions over up to a 22-day period.

The sixth part of this study will involve (a) subjects with previously diagnosed gingivitis, including moderate gingival inflammation (Löe and Silness Gingival Index ≥2) and pocket depths <4, and (b) subjects with previously diagnosed gingivitis (moderate gingival inflammation (Löe and Silness Gingival Index ≥2)) AND periodontitis including gingival bleeding, gingival inflammation, and at least four sites with probing pocket depths >4mm. Subjects will be randomly assigned to brush twice daily for up to 6 months with the test or the control dental gel. On Days 0, 30, 90, and 180, plaque levels (Quigley-Hein, Turesky Modification Plaque Index), gingival inflammation (Löe and Silness Gingival Index), gingival bleeding (modified Sulcus Bleeding Index) and periodontal pocket depths will be determined by one blinded, investigator (Dr. Wilder-Smith) using a periodontal probe. In vivo Optical Coherence Tomography (OCT) and Multiphoton Microscopy (MPM) may be used for in situ imaging if gingival/periodontitis sites are accessible to the imaging probes. The results from this study will help evaluate the effects of the test dentifrice formulation on plaque removal and maintaining/recovering gingival/periodontal health.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18
* Have a previously diagnosed condition of gingivitis and periodontitis including gingival bleeding, gingival inflammation, plaque, and for some study sections at least four sites with probing pocket depths > 4mm.
* Not pregnant and not lactating.

Exclusion Criteria:

* Participated in other clinical study within the last 30 days.
* Plan to receive dental treatment during the study dates.
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouth rinses.
* Allergies to personal care/consumer products or their ingredients.
* Less than 20 teeth (excluding third molars).
* For some studies, within six months prior to baseline, any quadrant or maintenance S/RP, and/or periodontal surgical therapy
* Diagnosed with active acquired immunodeficiency syndrome (AIDS) or Hepatitis B/C and other significant disease or disorder.
* Poorly controlled diabetes
* History of herpetic infection, recurrent aphthous ulcer, or other ulcerative diseases, abscesses, granulomas.
* History of or currently undergoing immunosuppression
* Taken antibiotics in the previous 3 months.
* Taking anti-inflammatory medications or Immunosuppressants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be recruited from University of California Irvine faculty, staff and students as well as individuals residing or working in the UCI neighborhood.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2014-10; Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Gingival health measure 1 | Up to 6 months
  Gingival Index
Gingival health measure 2 | Up to 6 months
  Sulcus Bleeding Index
Gingival health measure 3 | Up to 6 months
  Optical Coherence Tomography
Periodontal health measure 1 | Up to 6 months
  Optical Coherence Tomography
Periodontal health measure 2 | Up to 6 months
  Periodontal Pocket Depths
Plaque removal and reaccumulation measure 1 | Up to 6 months
  Plaque Index
Plaque removal and reaccumulation measure 2 | Up to 6 months
  Optical Coherence Tomography
Plaque removal and reaccumulation measure 3 | Up to 6 months
  Multiphoton microscopy

SECONDARY OUTCOMES:
Plaque characterization | Up to 6 months
  Multiphoton microscopy
Enamel health measure 1 | Up to 6 months
  SEM
Enamel health measure 2 | Up to 6 months
  microhardness
Enamel health measure 3 | Up to 6 months
  microCT
Enamel health measure 4 | Up to 6 months
  EDS
Enamel health measure 5 | Up to 6 months
  XPS

CONTACTS AND LOCATIONS:
Overall Officials: Petra Wilder-Smith, DDS, DMD, PhD, Principal Investigator — Beckman Laser Institute, UCI
Locations (1):
- Beckman Laser Institute, University of california, Irvine, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No